CLINICAL TRIAL: NCT00540683
Title: Measurement of the Distribution of Optical Properties in Adult Human Muscle
Status: Withdrawn | Type: Observational
Why Stopped: Not NIH defined clinical trials.
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Bruce Tromberg,Ph.D.,Director, Beckman Laser Institute and Medical Clinic and Professor, Departments of Biomedical Engineering and Surgery, University of California, Irvine
Other Study IDs: 20043626
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Muscle Disorder
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Diffuse Optical Spectroscopy — Muscle properties

SUMMARY:
The researcher can use Diffuse Optical spectroscopy technique that uses harmless levels of near-infrared light to probe the concentrations and states of important physiological molecules such as hemoglobin water and lipids in human muscle,.

DETAILED DESCRIPTION:
The researcher can monitor muscle physiology, for example during exercise or in response to external factors such as shock by Diffuse Optical spectroscopy technique.

The Diffuse Optical spectroscopy technique can determine significant changes in muscle, muscle structure, muscle tissues metabolism and hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 18 years and older
* Diagnosed of Cachexic condition
* Diagnosed of Cellulite adult female 18 years and older

Exclusion Criteria:

* Pregnant women
* Taking light sensitive drugs for use in photodynamic therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from outpatient clinic at University Of California Irvine, and staffs and students.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2004-10; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Healthy Muscle | upto 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Tromberg, Ph.D, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Beckman Laser Institute University of California Irvine, Irvine, California, United States